CLINICAL TRIAL: NCT04960930
Title: A Phase 3, Multi-center, Randomized, Double-Blind, Vehicle-controlled Study to Evaluate the Efficacy and Safety of Topical Administration of Minocycline Hydrochloride Foam (4%) in the Treatment of Moderate-to-Severe Acne Vulgaris
Brief Title: To Evaluate the Efficacy and Safety of Minocycline Hydrochloride Foam in the Treatment of Moderate-to-severe Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cutia Therapeutics (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CU-10201-301
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Drug: FMX101 FMX101, 4% minocycline foam
  Drug: Vehicle Foam Vehicle Foam
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMX101 (Experimental): FMX101 4% minocycline foam
  Interventions: Drug: FMX101
- Vehicle Foam (Placebo Comparator): Vehicle Foam
  Interventions: Drug: FMX101

INTERVENTIONS:
Drug: FMX101 — topically once daily

SUMMARY:
This is a randomized, multicenter, double-blind, vehicle-controlled, 2-arm study to evaluate the safety and efficacy in 12 weeks of FMX101 minocycline foam, 4%, compared to vehicle, in the treatment of subjects with moderate to severe facial acne vulgaris.

DETAILED DESCRIPTION:
Qualified subjects will be randomized to receive 1 of the following 2 treatments:

* FMX101 4% minocycline foam
* Vehicle foam

Subjects with qualifying lesion counts and Investigator's Global Assessments (IGA) of acne severity scores and will be assigned to 1 of 2 treatments according to the randomization schedule. Subjects will apply the assigned study drug topically once daily for 12 weeks as directed. Subjects will be advised to apply the study drug at approximately the same time each day, preferably in the evening at bedtime. Both the Investigator and subject will be blinded to the study drug identity.

Subjects will return for visits at Weeks 1, 2, 4, 6, 8, and 12. At the discretion of the clinic staff, for the convenience of subjects or clinic staff, visits can be scheduled to occur 2 days before or after the nominal schedule date for the Weeks 1, 2, 4, 8 and 12 visits. Efficacy evaluations (acne lesion counts and IGAs) will be performed at each visit during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Has completed and signed an appropriately administered Informed Consent Form (ICF) prior to any study-related procedures. Subjects less than 18 years of age (or as required by state law) must sign an Assent Form for the study and a parent or legal guardian must sign the ICF.
2. Has facial acne vulgaris with:

   * 20 to 50 inflammatory lesions (papules, pustules, and nodules)
   * 25 to 100 non-inflammatory lesions (open and closed comedones)
   * No more than 2 nodules on the face
   * IGA score of moderate (3) to severe (4)
3. Willing to use only the supplied non-medicated cleanser (Cetaphil Gentle Skin Cleanser) and to refrain from use of any other acne medication, medicated cleanser, excessive sun exposure, and tanning booths for the duration of the study.

Exclusion Criteria:

1. Acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne), or any dermatological condition of the face or facial hair (eg, beard, sideburns, mustache) that could interfere with the clinical evaluations.
2. Sunburn on the face.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
ILC | Week12
  The efficacy assessments will inflammation lesion counts at week12

SECONDARY OUTCOMES:
Investigator Global Assessment (IGA) | week 12
  Severity of acne vulgaris assessed by Investigator Global Assessment (IGA) IGA Scale for Acne Vulgaris for study is 0-5, score 0 is clear and normal, and score 5 is very severe.
nILC | week 12
  The efficacy assessments will non-inflammation lesion counts at baseline and week12
ILC week4 | week 4
  The Absolute Change From Baseline in the Inflammatory Lesion Count at Week 4
ILC week8 | week 8
  The Absolute Change From Baseline in the Inflammatory Lesion Count at Week 8
Investigator Global Assessment (IGA) week4 | Week 4
  IGA Treatment Success at Week 4 IGA Scale for Acne Vulgaris for study is 0-5, score 0 is clear and normal, and score 5 is very severe.
Investigator Global Assessment (IGA) week8 | Week 8
  IGA Treatment Success at Week 8 IGA Scale for Acne Vulgaris for study is 0-5, score 0 is clear and normal, and score 5 is very severe.

CONTACTS AND LOCATIONS:
Locations (29):
- China (29):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijin, Beijin
  - Beijing Tsinghua Changgung Hospital, Beijin, Beijin
  - The Southwest Hospital Of Amu, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Dermatology Hosptial of Southern Medical University, Yuexiu, Guangdong
  - The Second Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Xiangya Hospital Of Central South University, Changsha, Hunan
  - Institute of Dermatology Chinese Academy of Medical Sciences, Nanjin, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The First Bethune Hosptial of Jilin University, Changchun, Jiling
  - The First Hosptial of China Medical University, Shenyang, Liaoning
  - Shengjin Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hosptial of Qingdao University, Qingdao, Shandong
  - Shanghai Medical College of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital Skin Disease Hospital of Tongji University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjing, Tianjing
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hosptial Zhejiang University School Of Medicine, Hangzhou, Zhejiang